CLINICAL TRIAL: NCT07224165
Title: Developing a Digital Intervention for Adolescent Nonsuicidal Self-injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kaylee Kruzan, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STU00219136; K01MH131898 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Nonsuicidal Self-injury; Depression; Anxiety
MeSH Terms: conditions — Self-Injurious Behavior; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-guided digital intervention for NSSI (Experimental): This is the experimental condition
  Interventions: Device: App-based digital mental health intervention for adolescent NSSI
- Self-guided delivery of healthy living psychoeducational materials (Active Comparator): This is the comparison condition
  Interventions: Device: App-based delivery of healthy living psychoeducational materials

INTERVENTIONS:
Device: App-based digital mental health intervention for adolescent NSSI — The digital intervention for NSSI is an app-based intervention consisting of 16 modules (8 focused on internal skills and 8 focused on external sources of support) to be delivered twice weekly for 8 weeks. Modules containing psychoeducation and skill-based practice, and brief assessments. All content is delivered by a highly interactive conversational agent that guides users through the app content via a text-like interface. Psychoeducational content and strategies center on cognitive behavioral principles and support increased knowledge of external sources of support. Brief assessments examine NSSI and use of skills.
  Arms: Self-guided digital intervention for NSSI
Device: App-based delivery of healthy living psychoeducational materials — The control intervention is an app-based adolescent healthy living intervention consisting of 16 modules containing psychoeducation (e.g., sleep hygiene, water intake, exercise). Modifications will be made to an existing intervention used as a control in prior studies, 1,2 to mitigate potential contraindication for participants with eating disorder comorbidity by replacing nutrition with sun exposure content and an expansion of module content on sleep hygiene and exercise. Like the treatment app, all content in the control app is delivered by a highly interactive conversational agent that guides users through the app content via a text-like interface. Psychoeducational content and psychological strategies delivered center on stress management and healthy living.
  Arms: Self-guided delivery of healthy living psychoeducational materials

SUMMARY:
This is a feasibility trial of a digital mental health intervention aimed at adolescents (ages 14-18) with nonsuicidal self-injury and who are not currently engaged in mental health treatment. The study has two arms: a self-guided DMHI and an active control which will involve the delivery of non-interactive psychoeducational content via the same app interface. The primary goals of this project are to evaluate the feasibility of the intervention and trial procedures in preparation for a fully-powered randomized-controlled trial.

DETAILED DESCRIPTION:
The primary purpose of this trial is to test the feasibility of conducting a randomized controlled trial (RCT) of an 8-week digital mental health intervention (DMHI) for non-treatment engaged adolescents who engage in nonsuicidal self-injury. The DMHI will include a highly interactive conversational agent that conveys psychoeducational content and guides participants through skill-based activities. The study team will conduct a 2-arm feasibility trial, randomizing participants to receive either DMHI (weeks 1-8) or an active psychoeducational control (weeks 1-8). Participants will be 1:1 randomized to arms in varying block sizes of 4 and 6. To prevent allocation bias, randomization will be conducted by the biostatistician, who will not inform the study team of the treatment arms until the baseline assessment has been completed and the participant has been enrolled.

The primary clinical outcome measures will be frequency and severity of NSSI behavior (ABASI) and help-seeking activities (AHSQ). Implementation potential outcomes include intervention acceptability (IAM) and appropriateness (AIM).

This study will enroll individuals who have meet the following eligibility criteria: 1) Current NSSI, defined as NSSI on 2 or more days in the past month, as assessed by the Alexian Brothers Assessment of Self-Injury (ABASI). 2) English language skills sufficient to engage in the consent and intervention procedures. 3) Age 14 to 18. 4) Access to smartphone.

Exclusion criteria include: 1) Severe mental health diagnoses for which this intervention would be inappropriate (e.g., psychotic disorders, active manic episodes), 2) Severe suicide risk, including suicidal ideation with a plan and intent to act or history of suicide attempt in the past 3 months; or 3) Current engagement in psychotherapy (at baseline and for the trial recruitment only). Participants will be permitted to seek treatment at any point once enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Current NSSI (NSSI on 2 or more days in the last month
* English language skills sufficient to engage in the consent and intervention procedures
* Age 14-18
* Access to smartphone

Exclusion Criteria:

* Severe mental health diagnoses for which this intervention would be inappropriate (psychotic disorders, active manic episodes)
* Severe suicide risk, including suicidal ideation with a plan and intent to act
* Current engagement in psychotherapy

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Actual help-seeking questionnaire (AHSQ) | 16 weeks
  10-item measure assessing recent help-seeking from a variety of formal and informal sources
Alexian Brothers Assessment of Self-Injury - Methods checklist | 16 weeks
  16-item checklist that assesses the frequency (days/times) of common NSSI methods within the past month.
Acceptability of Intervention Measure (AIM) | 8 weeks
  4-item measure of intervention acceptability. Item responses are measured on a Likert scale from 1-5. So total scores can vary from 4-20 with 20 representing more acceptability.
Intervention Appropriateness Measure (IAM) | 8 weeks
  4-item measure of intervention appropriateness. Item responses are measured on a Likert scale from 1-5. So total scores can vary from 4-20 with 20 representing more appropriateness.

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through and managed by the NIMH Data Archive (NDA). De-identified human subjects data, harmonized to a common standard, are available to qualified researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available after publication of the primary outcome papers.
Access Criteria: The NIMH Data Archive is managed by the NIMH. Access criteria are determined by the NIMH.